CLINICAL TRIAL: NCT04123561
Title: A Phase 3, Randomized, Double-blind, Placebo- and Active-controlled Study to Evaluate the Efficacy and Safety of TLC599 in Patients With Osteoarthritis of the Knee
Brief Title: Extended and Controlled Release Liposomal Formulated Dexamethasone for Chronic Knee OA Pain
Acronym: EXCELLENCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taiwan Liposome Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TLC599A3005
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — dexamethasone 21-phosphate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TLC599 (Experimental): TLC599 (1mL) IA injection
  Interventions: Drug: TLC599
- Dexamethasone sodium phosphate (Active Comparator): DSP 4mg (1mL) IA injection
  Interventions: Drug: TLC599; Drug: DSP
- Normal Saline (Placebo Comparator): Normal saline (1mL) IA injection
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: TLC599 — TLC599 is a proprietary (Bioseizer) lipid formulation containing DSP (active ingredient)
  Other Names: TLC599 Injection
  Arms: Dexamethasone sodium phosphate; TLC599
Drug: DSP — Dexamethasone sodium phosphate (DSP) is a glucocorticoid widely used in the treatment of joint pain such as gout, osteoarthritis and rheumatoid arthritis via IA injection.
  Other Names: Dexamethasone Sodium Phosphate
  Arms: Dexamethasone sodium phosphate
Other: Normal Saline — 0.9% normal saline
  Arms: Normal Saline

SUMMARY:
Phase 3 randomized, double-blind, placebo- and active comparator-controlled study of TLC599.

DETAILED DESCRIPTION:
This is a Phase 3 randomized, double-blind, placebo- and active comparator-controlled pivotal study. Approximately 500 adult patients with moderate to severe pain due to OA of the knee will be enrolled and randomized. All patients will be followed for a total of 52 weeks. Efficacy and safety of 2 doses of TLC599 will be evaluated in comparison to Placebo and DSP through Week 52.

ELIGIBILITY:
Inclusion Criteria:

Male or female ≥40 years of age. BMI ≤ 40 kg/m2. Radiographically documented OA with Kellgren-Lawrence severity Grade 2 or 3 and associated symptoms Patient-reported pain with NRS score ≥4 (on a 0-10 scale) Able to read, understand, and sign the informed consent form, communicate with the investigator, complete study diaries, and understand and comply with protocol requirements.

Exclusion Criteria:

Recent use of IA or systemic corticosteroids Patient who is not ambulatory Any surgery or arthroscopy in the index knee within 12 months Any condition that could possibly confound the patient's assessment of index knee pain Substance abuse disorder, or positive urine drug test for illegal drug substances History of acquired or congenital immunodeficiency diseases History of treated malignancy which is disease free for ≤5 years Known allergy or hypersensitivity to the study drugs or their components

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Brown, PhD, Study Director — Taiwan Liposome Company
Locations (46):
- United States (41):
  - Cahaba Research, Inc, Birmingham, Alabama
  - Affinity Orthopedic Specialists Llc, Birmingham, Alabama
  - Shoals Medical Trials Inc, Sheffield, Alabama
  - Gb Family Care, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Clinical Research Institute of Arizona Llc, Surprise, Arizona
  - Noble Clinical Research Llc, Tucson, Arizona
  - Biosolutions Clinical Research Center, La Mesa, California
  - Translational Reseach Group Inc Dba Providence Clinical Research, North Hollywood, California
  - Prospective Research Innovations Inc, Rancho Cucamonga, California
  - Encompass Clinical Research, Spring Valley, California
  - Chase Medical Research Llc, Waterbury, Connecticut
  - Tampa Bay Medical Research, Clearwater, Florida
  - University Clinical Research-Deland, Llc Dba Accel Clinical Research, DeLand, Florida
  - Jacksonville Center For Clinical Research, Jacksonville, Florida
  - Charter Research, Llc, Lady Lake, Florida
  - Well Pharma Medical Research Corp, Miami, Florida
  - Conquest Research, Llc, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Conquest Research (Winter Park), Winter Park, Florida
  - Drug Studies America, Marietta, Georgia
  - Georgia Institute For Clinical Research Llc, Marietta, Georgia
  - Better Health Clinical Research Inc, Newnan, Georgia
  - Chicago Clinical Research Institute, Inc., Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Healthcare Research Network Ii, Llc, Flossmoor, Illinois
  - Affinity Health, Oak Brook, Illinois
  - Medisphere Medical Research Center Llc, Evansville, Indiana
  - Professional Research Network of Kansas Llc, Wichita, Kansas
  - Delricht Research, New Orleans, Louisiana
  - Healthcare Research Network, Hazelwood, Missouri
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Drug Trials America, Hartsdale, New York
  - Lillestol Research Llc, Fargo, North Dakota
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Lowcountry Orthopedics C/O Coastal Carolina research center, North Charleston, South Carolina
  - Clinical Investigations of Texas, Plano, Texas
  - Quality Research Inc, San Antonio, Texas
  - Clinical Trials of Texas Inc (Ctt), San Antonio, Texas
  - Charlottesville Medical Research Center Llc, Charlottesville, Virginia
- Australia (5):
  - Genesis Research Services, Broadmeadow, New South Wales
  - Australian Clinical Research Network, Maroubra, New South Wales
  - Northern Sydney Local Health District, Saint Leonards, New South Wales
  - Austrials, Taringa, Queensland
  - Colin Bayliss Research and Teaching Unit, Victoria Park, Western Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened for study eligibility at multiple study centers in the United States (US) and Australia.
Groups:
- TLC599 12 mg: TLC599: 1 mL IA injection
  TLC599 is a proprietary (Bioseizer) lipid formulation containing DSP (active ingredient)
- DSP 4 mg: DSP 4 mg: 1 mL IA injection
  Dexamethasone sodium phosphate (DSP) is a glucocorticoid widely used in the treatment of joint pain such as gout, osteoarthritis and rheumatoid arthritis via IA injection.
- Placebo: Normal saline: 1 mL IA injection
Period: Overall Study
Arm/Group | TLC599 12 mg | DSP 4 mg | Placebo
Started | 252 | 126 | 126
Completed | 208 | 96 | 101
Not Completed | 44 | 30 | 25
Not completed — Lost to Follow-up | 20 | 12 | 5
Not completed — Withdrawal by Subject | 9 | 7 | 9
Not completed — Lack of Efficacy | 7 | 8 | 6
Not completed — Adverse Event | 5 | 2 | 3
Not completed — A surgical procedure or IA administration in the index knee | 3 | 0 | 1
Not completed — Death | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) includes all randomized patients who receive study drug at baseline.
Groups:
- TLC599 12 mg: TLC599:1 mL IA injection
  TLC599 is a proprietary (Bioseizer) lipid formulation containing DSP (active ingredient)
- DSP 4 mg: DSP 4mg:1 mL IA injection Dexamethasone sodium phosphate (DSP) is a glucocorticoid widely used in the treatment of joint pain such as gout, osteoarthritis and rheumatoid arthritis via IA injection.
- Total: Total of all reporting groups
Arm/Group | TLC599 12 mg | DSP 4 mg | Placebo | Total
Number analyzed (Participants) | 252 | 126 | 126 | 504
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 162 | 81 | 79 | 322
  >=65 years | 90 | 45 | 47 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (8.50) | 59.9 (9.50) | 61.3 (9.30) | 61.0 (8.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 71 | 79 | 296
  Male | 106 | 55 | 47 | 208
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 17 | 18 | 79
  Not Hispanic or Latino | 207 | 107 | 108 | 422
  Unknown or Not Reported | 1 | 2 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 3 | 4
  Asian | 8 | 5 | 5 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  Black or African American | 48 | 26 | 20 | 94
  White | 195 | 94 | 95 | 384
  More than one race | 0 | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 224 | 114 | 109 | 447
  Australia | 28 | 12 | 17 | 57
Mean body mass index [Mean (Standard Deviation); unit: kg/m^2] — Body measurements - Mean body mass index (Kg/m^2)
  kg/m^2 | 31.13 (4.772) | 31.80 (5.144) | 31.33 (4.603) | 31.35 (4.825)
Mean weight [Mean (Standard Deviation); unit: Kg] — Body measurements - Mean weight (kg)
  Kg | 89.30 (17.816) | 91.71 (19.425) | 89.55 (17.750) | 89.96 (18.207)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in WOMAC Pain at Week 12 for TLC599 12 mg Versus Placebo
Description: The WOMAC (Western Ontario & McMaster Universities Osteoarthritis Index, Version 3.1) consists of 24 questions rated on a 0-4 Likert scale, totaling a score from 0-96, reflecting the previous 24 hours. Sub-scale scores for Pain (5 items, a 0-20 scale), Stiffness (2 items, a 0-8 scale), and Physical Function (17 items, a 0-68 scale) are summed to calculate the WOMAC Composite score. Both composite and sub-scale scores are normalized to a 0-4 scale for analysis, with higher scores indicating greater severity.
Time Frame: Baseline, Week 12
Population: The Full Analysis Set (FAS) includes all randomized patients who receive study drug at baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- TLC599 12mg: TLC599 :1mL IA injection
  TLC599 is a proprietary (Bioseizer) lipid formulation containing DSP (active ingredient)
- Placebo: Normal saline: 1mL IA injection
Arm/Group | TLC599 12mg | Placebo
Number analyzed (Participants) | 252 | 126
score on a scale | -0.968 [-1.060 to -0.877] | -0.798 [-0.930 to -0.665]
Statistical Analysis 1: Comparison: TLC599 12mg vs Placebo; Test type: Superiority — The primary efficacy endpoint is defined as the change from Injection 1 Baseline in WOMAC Pain on a normalized scale of 0-4 at Week 12 between the randomized TLC599 12mg and Placebo groups. The least-squares mean, alongside its corresponding 95% confidence interval, was used to estimate the treatment difference between TLC599 and Placebo, utilizing two-sided p-values; p = 0.0372, ANCOVA; Parameters estimated via REML using the Newton-Raphson algorithm, and the Kenward-Roger method calculates denominator degrees of freedom; Least Squares Mean Difference (LSMD) = -0.171, 95% CI 2-sided [-0.331 to -0.010], Standard Error of Mean 0.0819

2. Secondary Outcome: Change From Baseline in WOMAC Pain at Week 16 for TLC599 12 mg Versus Placebo
Description: as for outcome 1
Time Frame: Baseline, Week 16
Population: The Full Analysis Set (FAS) includes all randomized patients who receive study drug at baseline.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | TLC599 12mg | Placebo
Number analyzed (Participants) | 252 | 126
score on a scale | -0.929 (0.0492) | -0.798 (0.0704)

3. Secondary Outcome: Change From Baseline in WOMAC Pain at Week 20 for TLC599 12 mg Versus Placebo
Description: as for outcome 1
Time Frame: Baseline, Week 20
Population: The Full Analysis Set (FAS) includes all randomized patients who receive study drug at baseline.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Normal Saline: Normal saline: 1mL IA injection
Arm/Group | TLC599 12mg | Normal Saline
Number analyzed (Participants) | 252 | 126
score on a scale | -0.873 (0.0489) | -0.749 (0.0703)

4. Secondary Outcome: Change From Baseline in WOMAC Pain at Week 24 for TLC599 12mg Versus Placebo
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: The Full Analysis Set (FAS) includes all randomized patients who receive study drug at baseline.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | TLC599 12mg | Placebo
Number analyzed (Participants) | 252 | 126
score on a scale | -0.845 (0.0496) | -0.688 (0.0719)

5. Secondary Outcome: Change From Baseline in WOMAC Pain at Week 36 for TLC599 12mg Versus Placebo
Description: as for outcome 1
Time Frame: Baseline, Week 36
Population: The Full Analysis Set (FAS) includes all randomized patients who receive study drug at baseline.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | TLC599 12mg | Placebo
Number analyzed (Participants) | 252 | 126
score on a scale | -0.964 (0.0545) | -0.882 (0.0791)

6. Secondary Outcome: Change From Baseline in WOMAC Function at Week 12 for TLC599 12mg Versus Placebo
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: The Full Analysis Set (FAS) includes all randomized patients who receive study drug at baseline.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | TLC599 12mg | Placebo
Number analyzed (Participants) | 252 | 126
score on a scale | -0.903 (0.0470) | -0.735 (0.0681)

7. Secondary Outcome: PGIC at Week 12 for TLC599 12mg Versus Placebo
Description: Patient Global Impression of Change (PGIC) is a single-item question that measures change in patients' overall improvement rated on a 7-point scale including "1 = very much improved," "2 = much improved," "3 = minimally improved," "4 = no change," "5 = minimally worse," "6 = much worse," or "7 = very much worse".
Time Frame: Week 12
Population: The Full Analysis Set (FAS) includes all randomized patients who receive study drug at baseline.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | TLC599 12mg | Placebo
Number analyzed (Participants) | 252 | 126
score on a scale | 2.554 (0.0739) | 2.791 (0.1059)

8. Secondary Outcome: Total Rescue Acetaminophen Consumption Through Week 12 for TLC599 12mg Versus Placebo
Description: Rescue medication use of acetaminophen was provided and recorded in electronic patient diaries. Weekly Total Acetaminophen consumption was tabulated for analysis on a weekly basis, starting from the first date of study drug injection: (Day 1, 8), (Day 8, 15), and so on. Average daily use (e.g., Weekly Total Acetaminophen Consumption divided by 7) was computed to produce Weekly Average Daily Acetaminophen Consumption.
Time Frame: through Week 12
Population: The Full Analysis Set (FAS) includes all randomized patients who receive study drug at baseline.
Measure: Least Squares Mean (Standard Error); unit: tablets per week
Arm/Group | TLC599 12mg | Placebo
Number analyzed (Participants) | 252 | 126
tablets per week | 15.568 (3.1902) | 29.803 (4.5893)

9. Secondary Outcome: Durable Responder With ≥30% Decrease in WOMAC Pain From Baseline for Weeks 4 Through 12 for TLC599 12mg Versus Placebo
Description: Durable responder endpoints were derived based on the imputed WOMAC pain data. A subject which has ≥ 30% decrease in pain response from Baseline at each visit within a specified time period (x-y). This was derived for patients based on the Injection 1 Baseline for the following time period (x-y): (4-12).
Time Frame: Weeks 4 through 12
Population: The Full Analysis Set (FAS) includes all randomized patients who receive study drug at baseline.
Measure: Number; unit: percentage of responder
Arm/Group | TLC599 12mg | Placebo
Number analyzed (Participants) | 252 | 126
percentage of responder | 45.5 | 39.0

10. Secondary Outcome: Change From Baseline in WOMAC Function at Week 36 for TLC599 12mg Versus Placebo
Description: as for outcome 1
Time Frame: Baseline, Week 36
Population: The Full Analysis Set (FAS) includes all randomized patients who receive study drug at baseline.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | TLC599 12mg | Placebo
Number analyzed (Participants) | 252 | 126
score on a scale | -0.907 (0.0540) | -0.787 (0.0774)

11. Secondary Outcome: PGIC at Week 36 for TLC599 12mg Versus Placebo
Description: as for outcome 7
Time Frame: Week 36
Population: The Full Analysis Set (FAS) includes all randomized patients who receive study drug at baseline.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- TLC599: TLC599 :1mL IA injection
  TLC599 is a proprietary (Bioseizer) lipid formulation containing DSP (active ingredient)
Arm/Group | TLC599 | Placebo
Number analyzed (Participants) | 252 | 126
score on a scale | 2.635 (0.0883) | 2.738 (0.1288)

12. Secondary Outcome: Change From Baseline in WOMAC Pain at Week 12 for TLC599 12mg Versus DSP 4 mg
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: The Full Analysis Set (FAS) includes all randomized patients who receive study drug at baseline.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- TLC599 12 mg: TLC599 :1mL IA injection
  TLC599 is a proprietary (Bioseizer) lipid formulation containing DSP (active ingredient)
- DSP 4 mg: Dexamethasone sodium phosphate (DSP) is a glucocorticoid widely used in the treatment of joint pain such as gout, osteoarthritis and rheumatoid arthritis via IA injection.
Arm/Group | TLC599 12 mg | DSP 4 mg
Number analyzed (Participants) | 252 | 126
score on a scale | -0.968 (0.0467) | -0.933 (0.0667)

13. Secondary Outcome: Change From Baseline in WOMAC Pain at Week 52 for TLC599 12mg Versus Placebo
Description: as for outcome 1
Time Frame: Baseline, Week 52
Population: The Full Analysis Set (FAS) includes all randomized patients who receive study drug at baseline.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | TLC599 12mg | Placebo
Number analyzed (Participants) | 252 | 126
score on a scale | -0.928 (0.0580) | -0.934 (0.0820)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signs the ICF through the end of the study. The AE collected duration will be up to 56 weeks, including a Screening period of up to 4 weeks before randomization, Injection 1 Period of 24 weeks and Injection 2 Period of 28 weeks.
Description: All adverse events (AEs) were coded using the MedDRA v23.1 terminology to classify corresponding MedDRA System organ class (SOC) and preferred term (PT) for standardization and summary purposes.
Groups:
- TLC599 12 mg: TLC599 :1 mL IA injection
  TLC599 is a proprietary (Bioseizer) lipid formulation containing DSP (active ingredient)
Arm/Group | TLC599 12 mg | DSP 4 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/252 | 0/126 | 1/126
Serious Adverse Events (participants affected / at risk) | 16/252 | 4/126 | 7/126
Other Adverse Events (participants affected / at risk) | 73/252 | 33/126 | 28/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TLC599 12 mg (N=252) | DSP 4 mg (N=126) | Placebo (N=126)
COVID-19 (Infections and infestations) | 4 (4) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hiatus hemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cerebral venous sinus thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
syncope (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TLC599 12 mg (N=252) | DSP 4 mg (N=126) | Placebo (N=126)
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 (35) | 5 (5) | 10 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (14) | 10 (10) | 1 (1)
COVID-19 (Infections and infestations) | 12 (12) | 8 (8) | 3 (3)
Urinary tract infection (Infections and infestations) | 9 (11) | 2 (2) | 7 (7)
Hypertension (Vascular disorders) | 9 (10) | 8 (8) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/61/NCT04123561/Prot_SAP_000.pdf